CLINICAL TRIAL: NCT03542851
Title: A Randomized, Placebo-Controlled, Double-Blind, Crossover Study of Oral BTD-001 in Adults With Idiopathic Hypersomnia
Brief Title: A Study of Oral BTD-001 in Adults With Idiopathic Hypersomnia
Acronym: ARISE2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Balance Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BTD-001 IH202
Record Dates: First submitted 2018-05-01; First posted 2018-05-31 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Idiopathic Hypersomnia
MeSH Terms: conditions — Idiopathic Hypersomnia | interventions — Pentylenetetrazole

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Subject Receives BTD001 first (Experimental)
  Interventions: Drug: Pentetrazol (PTZ); Drug: Placebo oral capsule
- Subject Receives Placebo first (Experimental)
  Interventions: Drug: Pentetrazol (PTZ); Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Pentetrazol (PTZ) — BTD-001 is an oral capsule of PTZ.
  Other Names: PTZ
Drug: Placebo oral capsule — Placebo will be presented as oral capsule.

SUMMARY:
This is a randomized, placebo-controlled, double-blind, crossover study of oral BTD-001 in adults with Idiopathic Hypersomnia.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, crossover study of oral BTD-001 in adults with Idiopathic Hypersomnia (IH). The objectives of this study are two-fold: 1) To evaluate the efficacy of BTD-001 in subjects with IH as reflected by changes in cognitive, sleep, functional, and quality-of-life measures and 2) To characterize the safety and tolerability of oral BTD-001 administered to subjects with IH.

ELIGIBILITY:
Inclusion Criteria:

* Males or Females age 18 to 70 years old
* Onset of hypersomnia between age 10 and 30 years of age
* An Epworth Sleepiness Scale score of greater than or equal to 11
* Able to comply with requirements for concomitant medications and consumption of caffeine, alcohol, tobacco and nicotine (if on stimulants, agree to adhere to stable regimen throughout the trial)
* Females with a negative pregnancy test AND who are non-lactating
* Sexually active females of childbearing potential must be willing to use a highly effective method of birth control
* Sexually active males must have a vasectomy or use condoms

Exclusion Criteria:

* History of any disorder causing hypersomnia other than IH
* Evidence of circadian-rhythm disorder
* Sleep apnea syndrome
* Use of CPAP
* Obese subjects with BMI greater than or equal to 35kg/m2
* History of or current seizure disorder or history of syncope, unexplained loss of consciousnesses or seizure in the past 3 years as well as any past history of benzodiazepine and/or barbiturate and/or alcohol-related withdrawal seizures
* Columbia-Suicide Severity Rating Scale (C-SSRS) findings consistent with significant history of or current suicidal ideation or behavior
* Subjects who fail to wash out medications for IH or any other prohibited medications
* Positive toxicology screen test during the Screening or Baseline Visits.
* Clinically significant abnormal findings from physical, electrocardiogram (ECG) or laboratory assessments at Screening
* History of or current significant pulmonary, cardiac, neurological or psychiatric disease, substance dependence, porphyria, malignancy (with exception of local cutaneous squamous or basal cell carinomas or local cervical squamous cell carcinoma resolved after resection) or hypothyroidism (unless euthyroid at Screening Visit and treated with a stable dose of medication for at least 3 months prior to the Baseline Visit).
* Participation in a clinical drug trial within 4 weeks of Screening Visit

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-05-29 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-28 (Estimated)

PRIMARY OUTCOMES:
The efficacy of BTD-001 in subjects with IH as reflected by the IH Symptom Diary | Change from baseline.
  Measurements: IH Symptom Diary.

SECONDARY OUTCOMES:
The efficacy of BTD-001 in subjects with IH as reflected by changes in functional measures. | Change from baseline.
  Measurements: ESS (Epworth Sleepiness Scale).
The efficacy of BTD-001 in subjects with IH as reflected by changes in sleep measures. | Change from baseline.
  Measurements: MWT (Maintenance of Wakefulness Test)

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Lam, Study Director — Chief Operating Officer
Locations (32):
- United States (32):
  - Sleep Disorders Center of Alabama, Birmingham, Alabama
  - Mayo Clinic Hospital, Scottsdale, Arizona
  - SDS Clinical Trials, Orange, California
  - Pacific Research Network, San Diego, California
  - Sleep Medicine Specialists of California, San Ramon, California
  - Santa Monica Clinical Trials, Santa Monica, California
  - REM Sleep Medicine, Boulder, Colorado
  - PAB Clinical Research, Brandon, Florida
  - Sleep Medicine Specialists of South Florida, Miami, Florida
  - Florida Premier Research Institute, Winter Park, Florida
  - NeuroTrials Research Inc., Atlanta, Georgia
  - Sleep Practicioners, Macon, Georgia
  - Northshore Sleep Medicine, Northbrook, Illinois
  - Fort Wayne Neurology, Fort Wayne, Indiana
  - Rowe Neurology Institute, Lenexa, Kansas
  - Kentucky Research Group, Louisville, Kentucky
  - The Center for Sleep and Wake Disorders, Chevy Chase, Maryland
  - NeuroCare, Newton, Massachusetts
  - Sleep and Attention Disorders Institute, Sterling Heights, Michigan
  - Neuroscience Center, Saint Paul, Minnesota
  - St. Luke's Sleep Medicine and Research Center, Chesterfield, Missouri
  - Columbia University - Department of Neurology, New York, New York
  - Albert Einstein College of Medicine, New York, New York
  - Research Carolina of Huntersville, Huntersville, North Carolina
  - Intrepid Research, Cincinnati, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Geisinger, Danville, Pennsylvania
  - Consolidated Clinical Trials, Monroeville, Pennsylvania
  - Bogan Sleep Consultants, LLC, Columbia, South Carolina
  - Future Search Trials, Austin, Texas
  - Houston Sleep Center, Houston, Texas
  - Swedish Medical Center, Seattle, Washington